CLINICAL TRIAL: NCT02247128
Title: Antiplatelet Therapy for Patients Undergoing Transcatheter Aortic Valve Implantation
Acronym: POPular-TAVI
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: St. Antonius Hospital (Other)
Responsible Party: Principal Investigator, J.M. ten Berg, Prof. Dr., St. Antonius Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: POPTAV006
Record Dates: First submitted 2014-09-19; First posted 2014-09-23 (Estimated); Last update posted 2020-04-30 (Actual); Status verified 2020-04

CONDITIONS: Aortic Valve Disease; Myocardial Infarction; Stroke; Bleeding
Keywords: Transcatheter Aortic Valve Implantation (TAVI); Transcatheter Aortic Valve Replacement (TAVR); Aortic Valve Disease; Aortic Stenosis; Myocardial Infarction; Ischemic stroke; Bleeding; Thrombosis; Myocardial Ischemia; Heart Diseases; Cardiovascular Diseases; Vascular Diseases; Embolism and Thrombosis; Aspirin; Clopidogrel; Prasugrel; Ticagrelor; Antithrombotic treatment; Oral anticoagulation; Warfarin; Platelet Aggregation Inhibitors; Genetic Testing; Cytochrome P450 2C19 (CYP2C19); Prostaglandin-endoperoxide synthase 2(PTGS2)
MeSH Terms: conditions — Aortic Valve Disease; Myocardial Infarction; Stroke; Hemorrhage; Aortic Valve Stenosis; Ischemic Stroke; Thrombosis; Myocardial Ischemia; Heart Diseases; Cardiovascular Diseases; Vascular Diseases; Embolism and Thrombosis | interventions — Aspirin; Clopidogrel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Aspirin + Clopicogrel (Cohort A) (Active Comparator): Cohort A: patients will receive clopidogrel (75mg quaque die (qD), 3 months) on top of low-dose aspirin (≤100mg qD, at least 1 year but recommended lifelong). When a patient in Cohort A doesn't already takes aspirin, a loading dose of 300mg will be given within 24 hours prior to TAVI. The loading dose for clopidogrel is 300mg, and will be given within 24 hours prior to TAVI.
  Interventions: Drug: Aspirin + clopidogrel
- Aspirin monotherapy (Cohort A) (Active Comparator): Cohort A: patients will receive low-dose aspirin (≤100mg qD, at least 1 year but recommended lifelong). When a patients doesn't already takes aspirin, a loading dose of 300mg will be given within 24 hours prior to TAVI. It is recommended to omit other antiplatelet therapy (e.g. clopidogrel) at least 5 days prior to the TAVI procedure.
  Interventions: Drug: Aspirin monotherapy
- OAC + Clopicogrel (Cohort B) (Active Comparator): Cohort B: patients will receive clopidogrel (75mg qD, 3 months) on top of OAC (according to its indication). The loading dose for clopidogrel is 300mg, and will be given within 24 hours prior to TAVI. It is recommended to omit other antiplatelet therapy (e.g. aspirin) at least 5 days prior to the TAVI procedure.
  Interventions: Drug: OAC + clopicogrel
- OAC monotherapy (Cohort B) (Active Comparator): Cohort B: patients will receive OAC according to its indication. It is recommended to continue the OAC therapy peri-procedural (International Normalized Ratio aimed at 2.0). It is recommended to omit antiplatelet therapy (e.g. clopidogrel) at least 5 days prior to the TAVI procedure.
  Interventions: Drug: OAC monotherapy

INTERVENTIONS:
Drug: Aspirin + clopidogrel
  Arms: Aspirin + Clopicogrel (Cohort A)
Drug: Aspirin monotherapy
  Arms: Aspirin monotherapy (Cohort A)
Drug: OAC + clopicogrel
  Arms: OAC + Clopicogrel (Cohort B)
Drug: OAC monotherapy
  Arms: OAC monotherapy (Cohort B)

SUMMARY:
At present, a variety of antithrombotic regimens are prescribed in the early postprocedure period after transcatheter aortic valve implantation (TAVI). Dual antiplatelet therapy (DAPT) using aspirin and a thienopyridine in the initial period after TAVI is the recommended strategy; however, mono antiplatelet therapy using aspirin is suggested not to be inferior. In patients with atrial fibrillation (AF) or another indication for oral anticoagulation (OAC), no recommendations on best treatment regimen currently exist although triple therapy (OAC + DAPT) is best avoided due to increased bleeding risk.

We hypothesise that the omission of clopidogrel in the first 3 months after TAVI is safer and not less beneficial than the addition of clopidogrel to aspirin (cohort A) or OAC (cohort B).

DETAILED DESCRIPTION:
The trial consists of two cohorts:

* Cohort A, patients without an indication for OAC prior to TAVI.
* Cohort B, patients with an indication for OAC prior to TAVI (eg. atrial fibrillation, mechanic mitral valve prosthesis).

ELIGIBILITY:
Inclusion Criteria:

* Cohort A

  1. Patient has provided written informed consent.
* Cohort B

  1. Need for long-term oral anticoagulation;
  2. Patient has provided written informed consent.

Exclusion Criteria:

* Cohort A

  1. Need for long-term oral anticoagulation;
  2. Drug-eluting stent implantation within 3 months prior to TAVI procedure;
  3. Bare-metal stent implantation within 1 month prior to TAVI procedure;
  4. Allergy or intolerance to aspirin or clopidogrel.
* Cohort B

  1. Drug-eluting stent implantation within 3 months prior to TAVI procedure;
  2. Bare-metal stent implantation within 1 month prior to TAVI procedure;
  3. Allergy or intolerance to (N)OAC or clopidogrel.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1016 (Actual)
Dates: Start 2014-01; Primary Completion 2020-03 (Actual); Study Completion 2020-04 (Actual)

PRIMARY OUTCOMES:
Safety endpoint | 1 year
  The primary outcome is a safety endpoint, defined as freedom of all bleeding complications at 1 year after TAVI. The co-primary outcome is the safety endpoint defined as freedom of non-procedure related bleeding complications at 1 year after TAVI. For the classification of bleeding complications the Bleeding Academic Research Consortium Definition for Bleeding (BARC) bleeding classification is primarily used according to the Valve Academic Research Consortium (VARC).

SECONDARY OUTCOMES:
Net-clinical benefit endpoint | 1 year
  The secondary outcome is a net-clinical benefit endpoint, defined as freedom of the non-hierarchical composite of cardiovascular mortality, non-procedure related bleeding, stroke, or myocardial infarction at 1 year after TAVI.
Efficacy endpoint | 1 year
  The co-secondary outcome is an efficacy endpoint, defined as freedom of the non-hierarchical composite of cardiovascular mortality, ischemic stroke, or myocardial infarction at 1 year after TAVI.

OTHER OUTCOMES:
Pharmacoeconomics endpoint | 1 year
  Outcome measure is quality-adjusted life years

CONTACTS AND LOCATIONS:
Overall Officials: Jurrien M ten Berg, PhD, MD, Principal Investigator — St. Antonius Hospital; Pieter R Stella, MD, PhD, Principal Investigator — University Medical Center Utrecht (UMCU)
Locations (17):
- Belgium (6):
  - Algemeen Stedelijk Ziekenhuis, Aalst
  - Onze Lieve Vrouwe Ziekenhuis, Aalst
  - Imelda Ziekenhuis, Bonheiden
  - Algemeen Ziekenhuis Sint Jan, Bruges
  - Ziekenhuis Oost-Limburg, Genk
  - Universitair Ziekenhuis Leuven, Leuven
- Charles university, Third Faculty of Medicine, Prague, Czechia
- National Institute Surgery Cardiaque Et De Cardiologie Interventionnelle, Luxembourg, Luxembourg
- Netherlands (9):
  - Academic Medical Centre (AMC), Amsterdam, North Holland
  - Isala Clinics, Zwolle, Overijssel
  - St. Antonius Hospital, Nieuwegein, Utrecht
  - Medisch Spectrum Twente, Enschede
  - University Medical Center, Groningen
  - Universitair Medisch Centrum Leiden, Leiden
  - Academic Hospital, Maastricht
  - Haga Ziekenhuis, The Hague
  - University Medical Center Utrecht (UMCU), Utrecht

REFERENCES:
- [Derived] Brouwer J, Nijenhuis VJ, Delewi R, Hermanides RS, Holvoet W, Dubois CLF, Frambach P, De Bruyne B, van Houwelingen GK, Van Der Heyden JAS, Tousek P, van der Kley F, Buysschaert I, Schotborgh CE, Ferdinande B, van der Harst P, Roosen J, Peper J, Thielen FWF, Veenstra L, Chan Pin Yin DRPP, Swaans MJ, Rensing BJWM, van 't Hof AWJ, Timmers L, Kelder JC, Stella PR, Baan J, Ten Berg JM. Aspirin with or without Clopidogrel after Transcatheter Aortic-Valve Implantation. N Engl J Med. 2020 Oct 8;383(15):1447-1457. doi: 10.1056/NEJMoa2017815. Epub 2020 Aug 30. PMID 32865376
- [Derived] Nijenhuis VJ, Brouwer J, Delewi R, Hermanides RS, Holvoet W, Dubois CLF, Frambach P, De Bruyne B, van Houwelingen GK, Van Der Heyden JAS, Tousek P, van der Kley F, Buysschaert I, Schotborgh CE, Ferdinande B, van der Harst P, Roosen J, Peper J, Thielen FWF, Veenstra L, Chan Pin Yin DRPP, Swaans MJ, Rensing BJWM, van 't Hof AWJ, Timmers L, Kelder JC, Stella PR, Baan J, Ten Berg JM. Anticoagulation with or without Clopidogrel after Transcatheter Aortic-Valve Implantation. N Engl J Med. 2020 Apr 30;382(18):1696-1707. doi: 10.1056/NEJMoa1915152. Epub 2020 Mar 29. PMID 32223116
- [Derived] Nijenhuis VJ, Bennaghmouch N, Hassell M, Baan J Jr, van Kuijk JP, Agostoni P, van 't Hof A, Kievit PC, Veenstra L, van der Harst P, van den Heuvel AF, den Heijer P, Kelder JC, Deneer VH, van der Kley F, Onorati F, Collet JP, Maisano F, Latib A, Huber K, Stella PR, Ten Berg JM. Rationale and design of POPular-TAVI: antiPlatelet therapy fOr Patients undergoing Transcatheter Aortic Valve Implantation. Am Heart J. 2016 Mar;173:77-85. doi: 10.1016/j.ahj.2015.11.008. Epub 2015 Dec 1. PMID 26920599